CLINICAL TRIAL: NCT02776657
Title: Non-Invasive Assessment of Intracoronary Thrombosis in Patients With Acute Coronary Syndrome and Chronic Stable Angina Using Magnetic Resonance Imaging.
Brief Title: Intracoronary Thrombus Detection by Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015/0421
Record Dates: First submitted 2016-04-27; First posted 2016-05-18 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Angina Pectoris; Angina, Stable; Angina, Unstable; Myocardial Infarction
MeSH Terms: conditions — Angina Pectoris; Angina, Stable; Angina, Unstable; Myocardial Infarction | interventions — Magnetic Resonance Spectroscopy; Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Stable Angina) (Active Comparator): 20 patients with stable angina planned to undergo elective coronary angiography will be recruited and each participant will undergo magnetic resonance imaging (MRI) prior to invasive coronary angiography. During the angiogram, Optical Coherence Tomography (OCT) may be used to identify thrombus within the coronary arteries.
  Interventions: Other: Magnetic Resonance Imaging; Device: Optical Coherence Tomography; Procedure: Invasive Coronary Angiography
- Cohort 2 (Acute Coronary Syndrome) (Active Comparator): 20 patients diagnosed with acute coronary syndrome will be recruited and each participant will undergo magnetic resonance imaging (MRI) prior to invasive coronary angiography. During the angiogram, Optical Coherence Tomography (OCT) may be used to identify thrombus within the coronary arteries. If thrombus is identified, participants will be asked to undergo a repeat MRI scan at one and three months.
  Interventions: Other: Magnetic Resonance Imaging; Device: Optical Coherence Tomography; Procedure: Invasive Coronary Angiography

INTERVENTIONS:
Other: Magnetic Resonance Imaging — Each participant will undergo at least one MRI scan. A small number will be asked to undergo repeat MRI scanning at one and three months following the initial scan.
Device: Optical Coherence Tomography — Participants may undergo Optical Coherence Tomography (OCT) during the angiogram procedure in order to detect thrombus within the coronary arteries.
Procedure: Invasive Coronary Angiography — This will be performed as part of usual care and does not constitute part of the research project.

SUMMARY:
This study involves the use of Magnetic Resonance Imaging (MRI) to determine whether blood clots can be identified within the blood vessels supplying blood to the heart in patients with angina and who have recently suffered a heart attack.

DETAILED DESCRIPTION:
The majority of heart attacks are caused as a result of small blood clots forming within the blood vessels supplying blood to the heart, obstructing blood flow to the heart muscle. Research has also shown that blood clots may form in the blood vessels of the heart without causing a heart attack. At present, blood clots may be identified by techniques used during invasive coronary angiography, but we wish to determine whether a non-invasive test (MRI scanning) can be used to detect small blood clots within the blood vessels supplying blood to the heart muscle.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Previously diagnosed coronary artery disease undergoing elective invasive angiography (Cohort 1) OR
* Admitted with Acute Coronary Syndrome (ACS) diagnosed by two of the following criteria;

  1. Elevation of cardiac biomarkers (high sensitivity troponin I greater than 34ng/l in men and 16ng/l in women).
  2. Symptoms of myocardial ischaemia
  3. Electrocardiogram (ECG) changes indicative of acute ischaemia (Cohort 2)
* Planned invasive coronary angiography

Exclusion Criteria:

* Contraindication or inability to undergo MRI scanning
* Renal failure (estimated glomerular filtration rate less than 30millilitres/minute)
* Undergoing Primary Percutaneous Coronary Intervention
* Ongoing myocardial ischaemia or dynamic ECG changes
* Inability to provide informed consent
* Known allergy to gadolinium based contrast
* Women who are pregnant, breastfeeding or of child-bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01-14 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Evidence of high intensity signals within the coronary arteries on T1 weighted magnetic resonance imaging. | Within 72 hours prior to angiography

SECONDARY OUTCOMES:
The correlation between high risk plaques as determined on MRI with culprit plaques on invasive angiography in patients with acute coronary syndrome (ACS). | Through study completion, an average of 1 year
Incidence of intracoronary thrombosis, as detected by magnetic resonance imaging, in patients with stable coronary artery disease. | Through study completion, an average of 1 year
The change in plaque signal intensity on magnetic resonance imaging at one month following acute coronary syndrome (ACS). | Baseline and 1 month
The change in plaque signal intensity on magnetic resonance imaging at three months following acute coronary syndrome (ACS). | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Mhairi K Doris, MBChB, Principal Investigator — University of Edinburgh/NHS Lothian; David E Newby, PhD, Study Director — University of Edinburgh/NHS Lothian